CLINICAL TRIAL: NCT00062114
Title: A Phase II Study To Evaluate The Safety And Efficacy Of Zevalin (IND # BB IND 4850) Therapeutic Regimen In Patients With Transformed CD20 + B-Cell Non-Hodgkin's Lymphoma
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab in Treating Patients With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50201; CALGB-50201; CDR0000304498 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab + yttrium Y 90 ibritumomab tiuxetan (Experimental): Patients receive rituximab IV followed within 4 hours by yttrium Y 90 ibritumomab tiuxetan IV (for imaging) over 10 minutes on day 1. Patients undergo 1 (or 2 if needed) imaging scan between days 2-5. In the absence of altered biodistribution, patients receive rituximab IV followed within 4 hours by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8.
  Patients are followed monthly for 3 months, every 3 months for 2 years, and then every 6 months for 2 years.
  Interventions: Biological: rituximab; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies such as yttrium Y 90 ibritumomab tiuxetan and rituximab can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells.

PURPOSE: This phase II trial is studying how well giving yttrium Y 90 ibritumomab tiuxetan together with rituximab works in treating patients with progressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of yttrium Y 90 ibritumomab tiuxetan and rituximab, in terms of overall response rate (complete, unconfirmed complete, and partial) and duration of response, in patients with transformed CD20+ B-cell non-Hodgkin's lymphoma.
* Determine the safety of this regimen in these patients.
* Determine the event-free survival and time to treatment progression in patients treated with this regimen.
* Determine the immunogenicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV followed within 4 hours by indium In 111 ibritumomab tiuxetan IV (for imaging) over 10 minutes on day 1. Patients undergo 1 (or 2 if needed) imaging scan between days 2-5. In the absence of altered biodistribution, patients receive rituximab IV followed within 4 hours by yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8.

Patients are followed monthly for 3 months, every 3 months for 2 years, and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transformed CD20+ B-cell non-Hodgkin's lymphoma (NHL)

  * Transformation defined as:

    * Progression to a more aggressive diffuse lymphoma, excluding conversion to a more aggressive grade of follicular lymphoma (e.g., WHO/REAL follicular center, large, grade III NHL)
  * Initial large cell follicular lymphoma must progress to a diffuse large cell lymphoma
  * De novo transformed NHL ineligible
* Requiring treatment as determined by any of the following characteristics:

  * An increase in overall tumor size
  * Presence of B symptoms
  * Presence of masses that are causing ongoing clinical symptomatology
* Must have less than 25% bone marrow involvement with lymphoma
* Must have received and either relapsed or failed to respond to prior therapy for initial low grade or follicular NHL
* Must have bidimensionally measurable disease defined as:

  * Greater than 2 cm OR 1.5 cm if 0.5 cm slices are used during spiral CT scan
  * Nonmeasurable disease includes any of the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural or pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses that are not confirmed and followed by imaging techniques
    * Cystic lesions
    * Lesions that are situated in a previously irradiated area
* No expected impairment in bone marrrow reserve meeting any of the following criteria:

  * Platelet count less than 150,000/mm^3
  * Hypocellular bone marrow (less than 15% cellularity)
  * Marked reduction in bone marrow precursors of one or more cell lines (e.g., granulocytic, megakaryocytic, or erythroid)
  * History of failed stem cell collection
* Patients with peritoneal invasion and/or ascites with positive cytology for lymphoma OR pleural invasion and/or effusion with positive cytology for lymphoma are eligible only if their effusion or ascites can be tapped dry

  * No significant remaining malignant effusion or ascites at the time of study drug administration
* No known meningeal lymphoma or known parenchymal CNS lymphoma NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* Absolute neutrophil count at least 1,500/mm^3
* Lymphocyte count no greater than 5,000/mm^3
* Platelet count at least 150,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL

Renal

* Creatinine no greater than 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study treatment
* HIV negative
* No other malignancy except nonmelanoma skin cancer unless patient has completed therapy and is considered to be at less than 30% risk of relapse
* No human anti-mouse antibody (HAMA) reactivity (patients with prior exposure to murine antibodies)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Radiotherapy
* At least 3 weeks since prior anticancer immunotherapy (6 weeks for rituximab) and recovered
* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)
* No prior myeloablative therapy with bone marrow transplantation or peripheral blood stem cell rescue

Chemotherapy

* See Biologic therapy
* At least 3 weeks since prior anticancer chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered

Endocrine therapy

* No concurrent systemic corticosteroids with either of the following dose schedules:

  * No greater than 50 mg of prednisone as a single dose (or equivalent)
  * No greater than 50 mg of prednisone per dose (or equivalent) for more than 6 doses

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior anticancer radiotherapy and recovered
* No prior radioimmunotherapy, including yttrium Y 90 ibritumomab tiuxetan
* No prior external beam radiotherapy to more than 25% of active bone marrow (involved field or regional)

Surgery

* At least 3 weeks since prior anticancer surgery and recovered
* More than 4 weeks since prior major surgery (other than diagnostic surgery)

Other

* At least 3 weeks since other prior anticancer therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2004-04; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Up to 4 years
Duration of response | Up to 4 years

SECONDARY OUTCOMES:
Complete response (CR), unconfirmed CR, and partial response | Up to 4 years
Event-free survival | Up to 4 years
Time to progression | Up to 4 years
Time to next lymphoma treatment | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C. Shea, MD, Study Chair — UNC Lineberger Comprehensive Cancer Center
Locations (94):
- United States (94):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - Frisbie Memorial Hospital, Rochester, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming